CLINICAL TRIAL: NCT00397696
Title: Evaluation of 5-[123I]-A-85380 and SPECT Imaging as a Marker of Nicotinic Receptor Density in the Brain of Parkinson Disease Subjects
Brief Title: Evaluation of 5-[123I]-A-85380 and SPECT Imaging in Individuals With Parkinsons Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Danna Jennings, MD, Principal Investigator, Institute for Neurodegenerative Disorders
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5-IA02
Record Dates: First submitted 2006-11-07; First posted 2006-11-09 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson; imaging; nicotinic receptors
MeSH Terms: conditions — Parkinson Disease | interventions — Iodine-123

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- [123I] 5-IA (Experimental): To assess [123I] 5IA and SPECT imaging
  Interventions: Drug: [123I] 5-IA

INTERVENTIONS:
Drug: [123I] 5-IA — All subjects will undergo written informed consent and a screening evaluation including baseline clinical laboratory testing, a baseline physical and neurological evaluation and baseline cognitive evaluations using the MMSE, the ANAM computerized cognitive battery, and other tests of executive function. All subjects will be evaluated with United Parkinson Disease Rating Scales (UPDRS) following an overnight withdrawal of anti-parkinson medication. Subjects will be asked to undergo an injection of [123I] 5-IA followed by SPECT imaging as described below. A second [123I] 5-IA and SPECT imaging study will be obtained for reliability testing between 2 weeks and 2 months following the initial [123I] 5IA imaging session.

SUMMARY:
The underlying goal of this study is to assess [123I] 5-IA and SPECT imaging as a tool to detect nicotinic receptor activity in the brain of PD patients. All study procedures will be conducted at the Institute for Neurodegenerative Disorders (IND) and Molecular NeuroImaging (MNI) in New Haven, CT. Approximately 10 patients with a diagnosis of PD without cognitive changes will be recruited to participate in this study. Patients will be eligible to participate if they have a diagnosis of PD of more than 2 years duration and have no significant cognitive changes.

DETAILED DESCRIPTION:
All subjects will undergo written informed consent and a screening evaluation including baseline clinical laboratory testing, a baseline physical and neurological evaluation and baseline cognitive evaluations using the MMSE, the ANAM computerized cognitive battery, and other tests of executive function. All subjects will be evaluated with United Parkinson Disease Rating Scales (UPDRS) following an overnight withdrawal of anti-parkinson medication. Subjects will be asked to undergo an injection of [123I] 5-IA followed by SPECT imaging as described below. A second [123I] 5-IA and SPECT imaging study will be obtained for reliability testing between 2 weeks and 2 months following the initial [123I] 5IA imaging session.

The primary imaging outcome measure will be VT', the equilibrium distribution volume in brain regions is determined from an MRI-directed region-of-interest (ROI) analysis. The baseline imaging VT' will be compared to the follow-up imaging study to the reliability of the nicotinic [123I] 5-IA imaging.

ELIGIBILITY:
Inclusion Criteria:

* The presence of idiopathic Parkinson disease
* A clear clinical response to dopaminergic therapy treatment
* Hoehn and Yahr Stages < 3;
* 2-7 year Duration from time of diagnosis.
* Mini-mental status exam score of >24,
* For females, non-child bearing potential or negative urine pregnancy test on day of [123I] 5-IA injection.

Exclusion Criteria:

* Secondary Parkinsonism;
* Nicotine dependence or use within the previous 12 months prior to enrollment;
* Treatment with Aricept (donepezil), Exelon (rivastigmine), Cognex (tacrine) within the past 30 days; treatment with medications that bind to the nicotinic receptor.
* Clinically significant clinical laboratory value and/or medical or psychiatric illness;
* Mini-mental status exam score of ≤24.
* The subject has evidence of clinically significant thyroid disease, gastrointestinal, cardiovascular, hepatic, renal, hematologic, neoplastic, endocrine, neurologic, immunodeficiency, pulmonary, or other medical or psychiatric disorder;
* The subject has received an investigational drug within 30 days of the screening visit;
* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-11; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Radiotracer uptake in cortical regions in PD relative to Healthy Control subjects | 2 years
  Does [123I] 5-IA demonstrate qualitatively decreased radiotracer uptake in cortical regions consistent with a reduction in nicotinic receptor density in PD patients relative to controls?

SECONDARY OUTCOMES:
Nicotinic receptor as a reliable measure | 2 years
  Is [123I] 5-IA a reliable measure of nicotinic receptors in Parkinson Disease?

CONTACTS AND LOCATIONS:
Overall Officials: John Seibyl, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States

REFERENCES:
- [Background] Pirozzolo FJ, Hansch EC, Mortimer JA, Webster DD, Kuskowski MA. Dementia in Parkinson disease: a neuropsychological analysis. Brain Cogn. 1982 Jan;1(1):71-83. doi: 10.1016/0278-2626(82)90007-0. PMID 6927555
- [Background] Hoehn MM, Yahr MD. Parkinsonism: onset, progression and mortality. Neurology. 1967 May;17(5):427-42. doi: 10.1212/wnl.17.5.427. No abstract available. PMID 6067254
- [Background] Seibyl JP, Marek KL, Quinlan D, Sheff K, Zoghbi S, Zea-Ponce Y, Baldwin RM, Fussell B, Smith EO, Charney DS, van Dyck C, et al. Decreased single-photon emission computed tomographic [123I]beta-CIT striatal uptake correlates with symptom severity in Parkinson's disease. Ann Neurol. 1995 Oct;38(4):589-98. doi: 10.1002/ana.410380407. PMID 7574455
- [Background] Seibyl JP. Imaging studies in movement disorders. Semin Nucl Med. 2003 Apr;33(2):105-13. doi: 10.1053/snuc.2003.127303. PMID 12756643
- [Background] Marek K, Jennings D, Seibyl J. Single-photon emission tomography and dopamine transporter imaging in Parkinson's disease. Adv Neurol. 2003;91:183-91. No abstract available. PMID 12442677
- [Background] Marek K, Jennings D, Seibyl J. Dopamine agonists and Parkinson's disease progression: what can we learn from neuroimaging studies. Ann Neurol. 2003;53 Suppl 3:S160-6; discussion S166-9. doi: 10.1002/ana.10486. No abstract available. PMID 12666107
- [Background] Louis M, Clarke PB. Effect of ventral tegmental 6-hydroxydopamine lesions on the locomotor stimulant action of nicotine in rats. Neuropharmacology. 1998 Dec;37(12):1503-13. doi: 10.1016/s0028-3908(98)00151-8. PMID 9886673
- [Background] Parain K, Hapdey C, Rousselet E, Marchand V, Dumery B, Hirsch EC. Cigarette smoke and nicotine protect dopaminergic neurons against the 1-methyl-4-phenyl-1,2,3,6-tetrahydropyridine Parkinsonian toxin. Brain Res. 2003 Sep 12;984(1-2):224-32. doi: 10.1016/s0006-8993(03)03195-0. PMID 12932857
- [Background] O'Neill MJ, Murray TK, Lakics V, Visanji NP, Duty S. The role of neuronal nicotinic acetylcholine receptors in acute and chronic neurodegeneration. Curr Drug Targets CNS Neurol Disord. 2002 Aug;1(4):399-411. doi: 10.2174/1568007023339166. PMID 12769612
- [Background] Gale C, Martyn C. Tobacco, coffee, and Parkinson's disease. BMJ. 2003 Mar 15;326(7389):561-2. doi: 10.1136/bmj.326.7389.561. No abstract available. PMID 12637374
- [Background] Quik M, Kulak JM. Nicotine and nicotinic receptors; relevance to Parkinson's disease. Neurotoxicology. 2002 Oct;23(4-5):581-94. doi: 10.1016/s0161-813x(02)00036-0. PMID 12428730
- [Background] Mitsuoka T, Kaseda Y, Yamashita H, Kohriyama T, Kawakami H, Nakamura S, Yamamura Y. Effects of nicotine chewing gum on UPDRS score and P300 in early-onset parkinsonism. Hiroshima J Med Sci. 2002 Mar;51(1):33-9. PMID 11999458
- [Background] Ross GW, Petrovitch H. Current evidence for neuroprotective effects of nicotine and caffeine against Parkinson's disease. Drugs Aging. 2001;18(11):797-806. doi: 10.2165/00002512-200118110-00001. PMID 11772120
- [Background] Kelton MC, Kahn HJ, Conrath CL, Newhouse PA. The effects of nicotine on Parkinson's disease. Brain Cogn. 2000 Jun-Aug;43(1-3):274-82. PMID 10857708
- [Background] Aubert I, Araujo DM, Cecyre D, Robitaille Y, Gauthier S, Quirion R. Comparative alterations of nicotinic and muscarinic binding sites in Alzheimer's and Parkinson's diseases. J Neurochem. 1992 Feb;58(2):529-41. doi: 10.1111/j.1471-4159.1992.tb09752.x. PMID 1729398
- [Background] Zoghbi SS, Tamagnan G, Fujita M, Baldwin RM, Al-Tikriti MS, Amici L, Seibyl JP, Innis RB. Measurement of plasma metabolites of (S)-5-[123I]iodo-3-(2-azetidinylmethoxy)pyridine (5-IA-85380), a nicotinic acetylcholine receptor imaging agent, in nonhuman primates. Nucl Med Biol. 2001 Jan;28(1):91-96. doi: 10.1016/S0969-8051(00)00188-8. PMID 11182569